CLINICAL TRIAL: NCT06362083
Title: Construction of a Clinical Urethral Stricture Database for a Prospective Longitudinal Cohort Study
Brief Title: Urethral Stricture Database
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 34-317 ex 21/22
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Urethral Stricture
Keywords: Reconstructive surgery; Quality of life; Perioperative Outcomes
MeSH Terms: conditions — Urethral Stricture | interventions — Surveys and Questionnaires; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires and data collection — It is a non-interventional, single-center, non-randomized, prospective observational study obtaining data and patient-reported outcomes.

SUMMARY:
Establishment of a clinical urethral stricture database for a prospective longitudinal cohort study.

DETAILED DESCRIPTION:
The aim is to establish a prospective clinical database of patients undergoing urethral surgery due to urethral stricture. In addition to pre-operative basic data, intraoperative and postoperative data, as well as follow-up data through questionnaires, are to be collected. The main objective is the prospective determination of success rates of the performed urethral surgeries in the short, medium, and long term. Furthermore, risk factors leading to failure (recurrence of urethral stricture) should be identified. Ultimately, the quality of life before and after urethral surgery is to be assessed in order to compare the applied procedures.

In today's reconstructive urethral surgery, there are few scientific surveys so far. Many of the applied techniques (therapy options) are based more on the experiences of individual surgeons than on a solid database, hence there are also different approaches. By evaluating prospective data and comparing individually applied surgical methods, the least complication-prone and most successful techniques are to be identified. The planned study aims to create an "efficacy-safety" profile for each urethral surgery technique. This will enable us in the future to not only provide improved (data-based) patient information but also to involve the patient better in the therapy decision. Thus, in the future, counseling and therapy for a young sexually active patient could differ from counseling for an older patient who is no longer sexually active, even with the same stricture length and location.

The analyses of the urethral database will thus enable us to internally validate therapy algorithms and provide personalized patient counseling.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing any of the following urethral surgeries are included:

* Internal urethrotomy according to Sachse (endoscopic transurethral urethrotomy)
* End-to-end anastomosis
* Urethral plastic surgeries with oral mucosa graft (potentially penile skin)
* Urethral plastic surgeries with mesh graft
* Hypospadias corrections
* Boutonniere
* (Self) bougienage of the urethra

Exclusion Criteria:

* Lack of capacity to consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing urethral surgeries or interventions. All patients meeting the inclusion and exclusion criteria of the study should be informed about the possibility of participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2034-01-15 (Estimated); Study Completion 2034-03-15 (Estimated)

PRIMARY OUTCOMES:
Success rate of urethral reconstructive surgeries | Questionnaires to patients are captured 3, 6 an d12 months following surgery, and then every year put to 10 years
  Success is defined as a lack of stricture recurrence in the follow-up

SECONDARY OUTCOMES:
Complications of urethral reconstructive surgeries | Questionnaires to patients are captured 3, 6 an d12 months following surgery, and then every year put to 10 years
  Complications are defined as surgical site infection, fistula, problems at the preservation site of buccal mucosa.
Sexual function after urethral reconstructive surgeries | Questionnaires to patients are captured 3, 6 an d12 months following surgery, and then every year put to 10 years
Health status after urethral reconstructive surgeries | Questionnaires to patients are captured 3, 6 an d12 months following surgery, and then every year put to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Röthl Martina Anna, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No